CLINICAL TRIAL: NCT01759810
Title: Proteome-based Personalized Immunotherapy of Malignant Brain Tumors
Brief Title: Proteome-based Personalized Immunotherapy of Glioblastoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: NeuroVita Clinic (Other)
Collaborators: Blokhin's Russian Cancer Research Center (Other); Russian Foundation of Technological Development (Other); The Serbsky State Scientific Center for Social and Forensic Psychiatry (Other); National Institute of Regenerative Medicine (Other); SRC Bioclinicum (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBM/2012
Record Dates: First submitted 2012-12-28; First posted 2013-01-03 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Glioblastoma
Keywords: Glioblastoma, recurrent glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- allogeneic stem cells (Experimental): 3 ml suspension of allogeneic hematopoietic cells in 0.9%NaCl solution is administered in L3-L4 vertebrae interspace with 16-18G needle. The preparation is administered every 2 weeks for the first 2 months (at day 1, 14, 28, 42, 56). 2 ml of individual dendritic vaccine are administered subcutaneously in 4 points (shoulders and abdomen) 3 times every 14 days from the therapy beginning (at day 14, 28 and 42). Meloxicam, 7.5mcg once a day is started from day 7 till day 42. Preparation of cytotoxic lymphocytes is administered intrathecally once in 2 weeks during the first 3 months, and then once in a month for three months.
  Interventions: Biological: Dendritic vaccine, allogeneic hematopoietic stem cells, cytotoxic lymphocytes
- autologous stem cells (Active Comparator): 3 ml suspension of proteome-modified autologous hematopoietic cells in 0.9%NaCl solution is administered in L3-L4 vertebrae interspace with 16-18G needle. The preparation is administered every 2 weeks for the first 2 months (at day 1, 14, 28, 42, 56). 2 ml of individual dendritic vaccine are administered subcutaneously in 4 points (shoulders and abdomen) 3 times every 14 days from the therapy beginning (at day 14, 28 and 42). Meloxicam, 7.5mcg once a day is started from day 7 till day 42. Preparation of cytotoxic lymphocytes is administered intrathecally once in 2 weeks during the first 3 months, and then once in a month for three months.
  Interventions: Biological: Dendritic vaccine, autologous hematopoietic stem cells, cytotoxic lymphocytes

INTERVENTIONS:
Biological: Dendritic vaccine, allogeneic hematopoietic stem cells, cytotoxic lymphocytes
  Arms: allogeneic stem cells
Biological: Dendritic vaccine, autologous hematopoietic stem cells, cytotoxic lymphocytes
  Arms: autologous stem cells

SUMMARY:
Trial Hypothesis: Acute, progressing lethal neurooncological process can be transferred into chronic and non-lethal, the survival rates and life quality can be improved by of control of tumor cells (TCs) quantity and targeted regulation of effector functions of tumor stem cells (TSCs).

Brief Description:

The first line therapy of glioblastoma multiforme (GBM) involves allogeneic haploidentical hematopoietic stem cells (HSCs), dendritic vaccine (DV) and cytotoxic lymphocytes (CTLs).

TCs and TSCs are isolated from GBM sample. Dendritic cells are isolated from peripheral blood mononuclear cells and cultured. Tumor sample provides tumor specific antigens to prepare DV. CTLs are obtained from peripheral blood after DV administrations. HSCs are harvested from closely related donor after granulocyte-colony-stimulating factor (G-CSF) administration.

Allogeneic HSCs are administered intrathecally 5 times every 2 weeks, at day 1, 14, 28, 42, 56. DV is given 3 times every 2 weeks (day 14, 28, 42) subcutaneously in four points. CTLs are administered every 2 weeks for 3 months, then 3 times every 1 month intrathecally. Six months after the therapy completion, the efficiency is evaluated and the cohort demonstrating efficiency continues the therapy, while cohort demonstrating no efficiency is transferred to active comparator arm.

Second line therapy involves DV with recombinant proteins, CTLs and autologous HSC with modified proteome. Autologous HSCs are mobilized by G-CSF.

Carcinogenesis-free intracellular pathways of signal transduction able to respond to targeted regulation of therapeutic cell systems with specific properties, are detected in TSCs using complete transcriptome profiling of gene expression, proteome mapping and profiling of proteins, bioinformation and mathematical analysis and mathematical modeling of protein profiles. To find key oncospecific proteins in TSCs and TCs, the targets for TSCs regulation are detected, as well as protein ligands able to regulate reproductive and proliferative properties of TSCs.

Using these data of TCs and TSCs proteins, the cell preparations to initiate adoptive immune response are prepared: DV loaded with recombinant proteins analogous to key tumor antigens, CTLs and autologous proteome-modified HSCs.

Autologous proteome-modified HSCs, DV and CTLs are administered as in the first line therapy.

DETAILED DESCRIPTION:
The trial will include 60 cases of unresectable recurrent glioblastoma multiforme (GBM) after two lines of standard chemotherapy and complete course of radiotherapy.

The first line therapy of GBM involves allogeneic haploidentical hematopoietic stem cells (HSCs), dendritic vaccine (DV) and cytotoxic lymphocytes (CTLs).

HSCs are used to stimulate individualized adoptive immune response, to affect tumor cells (TCs) toxically and to regulate tumor stem cells (TSCs) targeted in order to suppress their reproductive and proliferative potential. To obtain HSC the donor receives 8 subcutaneous administrations of granulocyte colony-stimulating factor (G-CSF) with 8-10 hours interval for 4 days. The first three days a single dose is 2.5 mcg per 1 kg weight, the last day the dose is doubled. The stem cells are harvested at day 5. Red blood cells are withdrawn by centrifuging. The content of cell markers is evaluated by flow cytometry. The result is assessed after cytoconcentrate enrichment and removal of mature cells and plasma from it. The preparation is stored in tubes per 4 ml with cryoprotector and 10% polyglucin solution. Stem cell proportion is no less than 0.5x106 CD34+, and lymphocytes proportion is no less than 0.5x109 per one administration.

The sample of brain tumor is obtained through stereotaxic/ endoscopic/ open biopsy from all patients included into the trial. The TCs and TSCs are immunochemically isolated from GBM biopsy sample. One part of tumor sample is used for standard histological, cytological and immunochemical testing, while tumor cells (TCs) and tumor stem cells (TSCs) (CD133+) are isolated from the other part.

Dendritic cells are isolated from peripheral blood mononuclear cells and cultured. Tumor sample provides tumor specific antigens to prepare DV.

Preparation of CTLs aims to enhance cytotoxic effect on tumor due to great number of circulating CTLs. CTLs are isolated from about 100 ml of peripheral blood after 3 DV administrations, and of them dendritic cells (DCs) are grown. Then, peripheral blood is repeatedly taken, and lymphocytes are isolated. The CTLs are co-cultured with DCs loaded with tumor antigens (first line therapy) or recombinant proteins identical to key oncospecific proteins (second-line therapy) for several times to expand their number (108-109). Their immunophenotype is detected and CTLs are cryopreserved. The first stimulation of CTLs with DCs lasts 6-8 days, the second lasts 2-4 days, next 2 days the lymphocytes are stimulated for the third and fourth time. And then the received lymphocytes are stimulated by IL-2 for 2 days.

Six months after the first line therapy completion the efficiency is evaluated and the cohort demonstrating efficiency continues the therapy, while cohort demonstrating no efficiency will continue the trial with the second line therapy.

The second line therapy arm (active comparator arm) uses DV with recombinant proteins identical to key oncospecific proteins, autologous CTLs and autologous HSCs with modified proteome.

Autologous HSCs are received from the trial participant as described previously. Cell preparation of HSC for active comparator arm is obtained of the cytoconcentrate of autologous mononuclear cells of peripheral blood after mobilization as specified for experimental arm. Tumor specific antigens for active comparator group are provided by tumor tissue of the patient.

TCs and TSCs as well as HSCs of the patient undergo complete transcriptome mapping and gene expression profiling (CTMGEP) and proteome mapping and protein profiling (PMPP). Key (3 or 4 proteins with maximal normalized intensity) oncospecific proteins (OSP) are determined according to proteome testing of TCs, while proteome profiling of TSCs and use of databases of protein-protein relations permit detection of intracellular signal transduction pathways (ISTP) unaffected by carcinogenesis and capable of regulation. Also, receptor membrane targets to affect these signal pathways (acceptor membrane proteins) are detected, as well as proteins that are able to activate them (protein ligands). CTMGEP of TSCs confirms diagnosed functional ISTP. Mathematical modeling of CTMGEP and comparison with Affymetrix GeneChip Human genome U133A Array data reveals perturbagens able to chemically induce HSCs and to modify their proteome profile in order to provide secretion of requisite protein ligands. The database analysis permits understanding of how changes in gene expression induced by a low-molecular agent or micro RNA corresponds with the changes observed in the examined profile. If correspondence is significant, it is supposed, that the agent or similar agents can initiate the effect. If anticorrelation is significant, the agent is supposed to initiate an opposite effect in gene expression modification. The transcriptome of HSCs is modified by co-culturing mononuclear cells with perturbagens. Their biological efficiency is evaluated in vitro in Homunculus bioreactor. Then preparation is stored as described previously.

Individual DV is prepared from the leukoconcentrate of peripheral blood of the patient. The lymphocytes are isolated, cultured with G-CSF and interleukin-2, conditioned by tumor-specific antigens, TNF-α and PGE2 for 48 hours and loaded with recombinant proteins identical to key tumor-specific antigens detected at proteomic testing of TCs. Basic mechanism of individual DV immune effect is elaboration of tumor toxic lymphocytes by the organism of the patient.

CTLs are obtained as described previously. The intervention is described in the appropriate section.

Toxicity will be evaluated according to CTC-NCI criteria. Efficiency is assessed according to the following criteria:

1. Complete effect - -full disappearance of all tumor foci
2. Partial effect - -reduction of tumor size and/or metastatic foci by no less than 50% and no signs of new neoplasms
3. Stabilization - reduction of tumor foci size by less than 50% and no signs of new neoplasms
4. Progress - growth of tumor foci during the therapy. In case of mosaic effect, when part of foci progresses and part is stable or reducing, the therapy is continued but the cases are analyzed outside the context "Response to the therapy"

ELIGIBILITY:
Inclusion Criteria:

* Morphologically confirmed glioma (in case of relapse and impossibility of biopsy, diagnosis based on radiological and other diagnostic methods)
* Refractory to the first and following conventional lines of chemo- and radiotherapy, if their removal is impossible.
* Glioblastoma relapses after at least one line of conventional chemo- and radiotherapy, if their removal is impossible
* Availability of HLA partially compatible related donor
* Life expectancy of no less than 3 months
* Absence of severe decompensated organ dysfunction
* Informed consent of the patient or their parents
* Informed consent of the donor

Exclusion Criteria:

* Failure to meet one of the inclusion criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-12; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 2 years

SECONDARY OUTCOMES:
Complete disappearance of all tumor foci | 2 years

OTHER OUTCOMES:
reduction of tumor size by no less than 50% and absence of new foci | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrey S. Bryukhovetskiy, MD, Principal Investigator — ZAO "NeuroVita Clinic of Interventional and Restorative Neurology and Therapy"
Locations (1):
- ZAO "NeuroVita Clinic of Interventional and Restorative Neurology and Therapy", Moscow, Russia

REFERENCES:
- [Result] Bryukhovetskiy IS, Mischenko PV, Tolok EV, Zaitcev SV, Khotimchenko YS, Bryukhovetskiy AS. Directional migration of adult hematopoeitic progenitors to C6 glioma in vitro. Oncol Lett. 2015 Apr;9(4):1839-1844. doi: 10.3892/ol.2015.2952. Epub 2015 Feb 10. PMID 25789053
- [Result] Bryukhovetskiy A, Shevchenko V, Kovalev S, Chekhonin V, Baklaushev V, Bryukhovetskiy I, Zhukova M. To the novel paradigm of proteome-based cell therapy of tumors: through comparative proteome mapping of tumor stem cells and tissue-specific stem cells of humans. Cell Transplant. 2014;23 Suppl 1:S151-70. doi: 10.3727/096368914X684907. Epub 2014 Oct 9. PMID 25303679